CLINICAL TRIAL: NCT03293212
Title: Characteristics and Medical Resource Utilization of Postoperative Patients: A Cross-sectional Survey of Outpatients
Brief Title: Characteristics and Medical Resource Utilization of Postoperative Patients
Status: Completed | Type: Observational
Sponsor: Jaseng Medical Foundation (Other)
Collaborators: Korea Institute of Oriental Medicine (Other Government)
Responsible Party: Principal Investigator, In-Hyuk Ha, KMD, Director, Jaseng Medical Foundation
Other Study IDs: JS-CT-2017-03
Record Dates: First submitted 2017-09-19; First posted 2017-09-26 (Actual); Last update posted 2019-03-29 (Actual); Status verified 2018-02

CONDITIONS: Pain, Postoperative
Keywords: Postoperative pain; Failed back surgery syndrome; Korean medicine
MeSH Terms: conditions — Pain, Postoperative; Failed Back Surgery Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this study is to assess and analyze the characteristics and usage of conventional and Korean medical services in postoperative patients. This study therefore investigates the proportion of patients with a history of surgery out of patients visiting a spine-specialty Korean medicine hospital, and the prognosis and preference for conventional and Korean medicine treatment by previous treatment history in postoperative patients.

DETAILED DESCRIPTION:
A considerable number of patients suffer prolonged chronic pain that does not retract or diminish after surgery, and are thus unable to achieve the desired results in receiving surgical treatment. Postoperative pain is gradually being perceived as a social issue as opposed to a personal health condition. Meanwhile, although efforts to address chronic pain with integrative medicine are continued in answer to the lack of success of pain management through surgery, there is still a lack of supporting evidence.

The objective of this survey study is to assess the characteristics, usage of conventional and Korean medical services, and prognosis by period before and after surgery in postoperative patients visiting a Korean medicine hospital, and analyze the associations between the preference for conventional and Korean medicine treatment. This study therefore investigates the usage of conventional and Korean medical services in postoperative patients, and is expected to provide information that will potentially aid patient decision making.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chief complaint(s) of at least one or more of the following: low back pain (or radiating leg pain), neck pain (or radiating arm pain), knee pain, or shoulder pain
* Patients with a history of musculoskeletal surgery related to the chief complaint(s)
* Patients capable of effective communication with the researcher(s) and understanding the survey items
* Patients who have given written informed consent

Exclusion Criteria:

* Patients without a history of musculoskeletal surgery associated with the low back, neck, shoulder, or knee region(s)
* Patients whose current pain is mainly attributed to traffic accident injury
* Patients incapable of answering the researcher interviews and surveys
* Patients with other reasons rendering study participation inappropriate as judged by the researcher(s)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients newly visiting 4 sites of Jaseng Hospital of Korean Medicine due to postoperative pain
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2017-06-29 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2017-10-31 (Actual)

PRIMARY OUTCOMES:
Numeric rating scale (NRS) of pain | Within 7 days after 1st visit
  11-point pain scale

SECONDARY OUTCOMES:
Five level version of EuroQol-5 Dimension (EQ-5D-5L) | Within 7 days after 1st visit
  Health-related quality of life questionnaire consisting of 5 descriptive items and EQ Visual Analogue Scales (EQ-VASs)
Functional disability questionnaire (for low back pain patients as indicated by postoperative condition) | Within 7 days after 1st visit
  Oswestry Disability Index (ODI)
Functional disability questionnaire (for neck pain patients as indicated by postoperative condition) | Within 7 days after 1st visit
  Neck Disability Index (NDI)
Functional disability questionnaire (for knee pain patients as indicated by postoperative condition) | Within 7 days after 1st visit
  Western Ontario McMaster Universities Osteoarthritis Index (WOMAC)
Functional disability questionnaire (for shoulder pain patients as indicated by postoperative condition) | Within 7 days after 1st visit
  Shoulder Pain and Disability Index (SPADI)
Work Productivity and Activity Impairment Questionnaire: General Health (WPAI-GH) | Within 7 days after 1st visit
  Questionnaire assessing the effect of health problems on the ability to work and to perform regular activities
Beck Depression Inventory-II (BDI-II) | Within 7 days after 1st visit
  The Korean version of the BDI-II has been validated and consists of 21 multiple choice items for diagnosis of depression.
Medical service use | Within 7 days after 1st visit
  Type(s) of medical service use before and after surgery post-onset
Medical costs | Within 7 days after 1st visit
  Medical costs from medical service use before and after surgery post-onset
Satisfaction with and preference for conventional and Korean medicine | Within 7 days after 1st visit
  Satisfaction with and preference for conventional and Korean medicine as measured using a 9-point Likert scale

CONTACTS AND LOCATIONS:
Overall Officials: In-Hyuk Ha, KMD, M.Sc., Principal Investigator — Jaseng Medical Foundation
Locations (1):
- Jaseng Medical Foundation, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No